CLINICAL TRIAL: NCT02997943
Title: SMART Weight Loss Management
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: University of Michigan (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Bonnie Spring, Professor, Northwestern University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: NIH NIDDK R01DK108678; R01DK108678 (NIH)
Record Dates: First submitted 2016-12-05; First posted 2016-12-20 (Estimated); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Weight Loss
Keywords: Obesity; Weight Loss; Diet; Physical Activity; Mobile Health
MeSH Terms: conditions — Weight Loss; Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Step 1: Optimal First Line Treatment (Experimental): Participants will first be randomized to an optimal first line treatment in order to compare APP vs. APP + coaching. Participants assigned to Step 1 treatment "APP" will receive a study-specific smartphone application. Participants assigned to Step 1 treatment "APP + coaching" will receive a study-specific smartphone application plus 12 weekly telephone coaching sessions.
  Interventions: Behavioral: Step 1 Treatment: APP; Behavioral: Step 1 Treatment: APP + Coaching
- Step 2: Optimal Strategy to Address Nonresponse (Experimental): Beginning at week 2, participants who are identified as treatment non-responders will be re-randomized in order to compare two strategies to address non-response: a modest step-up or vigorous step-up treatment augmentation tactic. Step 2 treatment strategy: modest step-up will include provision of an additional mHealth intervention component (push notifications). Step 2 treatment strategy vigorous step-up will include provision of an additional mHealth intervention component (push notifications), plus a traditional weight loss intervention component (coaching, meal replacements). Participants will continue to receive their first line treatment.
  Interventions: Behavioral: Step 2 Treatment Strategy: Modest Step-up; Behavioral: Step 2 Treatment Strategy: Vigorous Step-up

INTERVENTIONS:
Behavioral: Step 1 Treatment: APP — Participants will receive a smartphone app to track weight, dietary intake and physical activity, and a technology core consisting of web-based weekly lessons, wireless scale, and activity tracker. Participants will use their own smartphone to receive the study smartphone application.
  Arms: Step 1: Optimal First Line Treatment
Behavioral: Step 1 Treatment: APP + Coaching — Participants will receive a smartphone app to track weight, dietary intake and physical activity; a technology core consisting of web-based weekly lessons, wireless scale, and activity tracker; 12 weekly telephone coaching sessions. Participants will use their own smartphone to receive the study smartphone application.
  Arms: Step 1: Optimal First Line Treatment
Behavioral: Step 2 Treatment Strategy: Modest Step-up — In addition to first line treatment, participants identified as non-responders will be provided an additional mHealth intervention component (push notifications) for the remaining 12 weeks.
  Arms: Step 2: Optimal Strategy to Address Nonresponse
Behavioral: Step 2 Treatment Strategy: Vigorous Step-up — In addition to the first line treatment, participants identified as non-responders will be provided an additional mHealth intervention component (push notifications) plus a traditional weight loss intervention component (coaching, meal replacements).
  Arms: Step 2: Optimal Strategy to Address Nonresponse

SUMMARY:
The overall objective of this study is to use an innovative experimental approach, the SMART (Sequential Multiple Assignment Randomized Trial), to determine the best way to sequence the delivery of mHealth tools and traditional treatment components in a stepped program of obesity treatments. The SMART approach is a highly efficient strategy for identifying and constructing efficacious adaptive interventions: it accommodates sequential decision-making based on the participant's response to early weight loss treatment components. The proposed treatment package begins with the least expensive components, and for participants identified as treatment non-responders, provides sequential step-up of additional treatment components. By sequentially delivering treatment components based on participant response, SMART permits achievement of the target outcome, weight loss, with least resource consumption and participant burden.

DETAILED DESCRIPTION:
The proposed study seeks to develop an effective, resource-sensitive strategy to manage weight loss treatment for obesity. During the 12-week active intervention phase, participants will be randomized to one of two first-line treatments: 1) mobile app alone (APP) or 2) app plus weekly telephone coaching sessions (APP+C). Beginning at week 2, those who are identified as treatment non-responders (did not lose an average of 0.5 lbs/week) will be re-randomized to one of two augmentation tactics: 1) Modest Step-up, operationalized as the addition of an additional mHealth component, or 2) Vigorous Step-up, operationalized as the addition of an additional mHealth component plus a traditional weight loss intervention component. Treatment responders will continue with the same first-line treatment. Treatment response be re-assessed at weeks 4 and 8. Those identified as treatment non-responders will be re-randomized at that time.

ELIGIBILITY:
Inclusion Criteria:

* 18 through 60 years old
* BMI between 27 - 45 kg/m2
* < 350 lbs
* Weight stable (no loss or gain >25 lbs. for the past 6 months)
* Interested in losing weight and not enrolled in a formal weight loss program or taking medications or supplements that may cause weight change
* Own a Smartphone and be willing to install the SMART App
* Reside in the Chicago area for the duration of their participation (12 months)

Exclusion Criteria:

* Unstable medical conditions (uncontrolled hypertension, diabetes - uncontrolled or treated with insulin, uncontrolled hypothyroidism, unstable angina pectoris, transient ischemic attack, cancer undergoing active treatment, cerebrovascular accident or myocardial infarction within the past six months, or Crohn's disease)
* Pregnancy, lactation, or intended pregnancy
* Active suicidal ideation, anorexia, bulimia, binge eating disorder, current substance abuse or dependence (besides nicotine dependence)
* Require assistive device for mobility or current condition that may limit or prevent participation in moderate activity
* Use of pacemaker or other electrical implanted device
* History of bariatric (or LapBand) surgery, or considering or currently on a wait-list for bariatric or LapBand surgery
* May not live with a current or past SMART study participant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2020-09-17 (Actual); Study Completion 2021-03-18 (Actual)

PRIMARY OUTCOMES:
Change in weight at 6 months | baseline, 6 months
  Weight measured in the lab, taken without shoes, wearing light clothing on a calibrated beam balance scale

OTHER OUTCOMES:
Change in weight at 12 months | baseline, 12 months
  Weight measured in the lab, taken without shoes, wearing light clothing on a calibrated beam balance scale
Cost effectiveness | 12 months
  Cost/pound lost of each study sequence embedded within the SMART design.

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Spring, PhD, Principal Investigator — Northwestern University; Inbal Nahum-Shani, PhD, Principal Investigator — University of Michigan
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pfammatter AF, Nahum-Shani I, DeZelar M, Scanlan L, McFadden HG, Siddique J, Hedeker D, Spring B. SMART: Study protocol for a sequential multiple assignment randomized controlled trial to optimize weight loss management. Contemp Clin Trials. 2019 Jul;82:36-45. doi: 10.1016/j.cct.2019.05.007. Epub 2019 May 23. PMID 31129369
- [Background] Nahum-Shani I, Smith SN, Spring BJ, Collins LM, Witkiewitz K, Tewari A, Murphy SA. Just-in-Time Adaptive Interventions (JITAIs) in Mobile Health: Key Components and Design Principles for Ongoing Health Behavior Support. Ann Behav Med. 2018 May 18;52(6):446-462. doi: 10.1007/s12160-016-9830-8. PMID 27663578
- [Background] Spring B, Pfammatter A, Alshurafa N. First Steps Into the Brave New Transdiscipline of Mobile Health. JAMA Cardiol. 2017 Jan 1;2(1):76-78. doi: 10.1001/jamacardio.2016.4440. No abstract available. PMID 27973672
- [Background] Spring B, Stump T, Penedo F, Pfammatter AF, Robinson JK. Toward a health-promoting system for cancer survivors: Patient and provider multiple behavior change. Health Psychol. 2019 Sep;38(9):840-850. doi: 10.1037/hea0000760. PMID 31436465
- [Background] Walton A, Nahum-Shani I, Crosby L, Klasnja P, Murphy S. Optimizing Digital Integrated Care via Micro-Randomized Trials. Clin Pharmacol Ther. 2018 Jul;104(1):53-58. doi: 10.1002/cpt.1079. Epub 2018 Apr 19. PMID 29604043
- [Background] Almirall D, Kasari C, McCaffrey DF, Nahum-Shani I. Developing Optimized Adaptive Interventions in Education. J Res Educ Eff. 2018;11(1):27-34. doi: 10.1080/19345747.2017.1407136. Epub 2017 Nov 29. PMID 29552270
- [Background] Wagner B 3rd, Liu E, Shaw SD, Iakovlev G, Zhou L, Harrington C, Abowd G, Yoon C, Kumar S, Murphy S, Spring B, Nahum-Shani I. ewrapper: Operationalizing engagement strategies in mHealth. Proc ACM Int Conf Ubiquitous Comput. 2017 Sep;2017:790-798. doi: 10.1145/3123024.3125612. PMID 29362728
- [Background] Welch WA, Spring B, Phillips SM, Siddique J. Moderating Effects of Weather-Related Factors on a Physical Activity Intervention. Am J Prev Med. 2018 May;54(5):e83-e89. doi: 10.1016/j.amepre.2018.01.025. Epub 2018 Mar 15. PMID 29551330
- [Background] Booth JN 3rd, Allen NB, Calhoun D, Carson AP, Deng L, Goff DC Jr, Redden DT, Reis JP, Shimbo D, Shikany JM, Sidney S, Spring B, Lewis CE, Muntner P. Racial Differences in Maintaining Optimal Health Behaviors Into Middle Age. Am J Prev Med. 2019 Mar;56(3):368-375. doi: 10.1016/j.amepre.2018.10.020. PMID 30777156
- [Background] Nahum-Shani I, Ertefaie A, Lu XL, Lynch KG, McKay JR, Oslin DW, Almirall D. A SMART data analysis method for constructing adaptive treatment strategies for substance use disorders. Addiction. 2017 May;112(5):901-909. doi: 10.1111/add.13743. Epub 2017 Feb 18. PMID 28029718
- [Background] Lu X, Nahum-Shani I, Kasari C, Lynch KG, Oslin DW, Pelham WE, Fabiano G, Almirall D. Comparing dynamic treatment regimes using repeated-measures outcomes: modeling considerations in SMART studies. Stat Med. 2016 May 10;35(10):1595-615. doi: 10.1002/sim.6819. Epub 2015 Dec 6. PMID 26638988
- [Background] Spring B, Champion KE, Acabchuk R, Hennessy EA. Self-regulatory behaviour change techniques in interventions to promote healthy eating, physical activity, or weight loss: a meta-review. Health Psychol Rev. 2021 Dec;15(4):508-539. doi: 10.1080/17437199.2020.1721310. Epub 2020 Feb 17. PMID 31973666
- [Background] Ertefaie A, Wu T, Lynch KG, Nahum-Shani I. Identifying a set that contains the best dynamic treatment regimes. Biostatistics. 2016 Jan;17(1):135-48. doi: 10.1093/biostatistics/kxv025. Epub 2015 Aug 3. PMID 26243172
- [Derived] Spring B, Pfammatter AF, Scanlan L, Daly E, Reading J, Battalio S, McFadden HG, Hedeker D, Siddique J, Nahum-Shani I. An Adaptive Behavioral Intervention for Weight Loss Management: A Randomized Clinical Trial. JAMA. 2024 Jul 2;332(1):21-30. doi: 10.1001/jama.2024.0821. PMID 38744428
- [Derived] Metzendorf MI, Wieland LS, Richter B. Mobile health (m-health) smartphone interventions for adolescents and adults with overweight or obesity. Cochrane Database Syst Rev. 2024 Feb 20;2(2):CD013591. doi: 10.1002/14651858.CD013591.pub2. PMID 38375882